CLINICAL TRIAL: NCT06099275
Title: Evaluation of Hemodynamics in People With Untreated Preeclampsia Using Echocardiography
Status: Suspended | Type: Observational
Why Stopped: inadequate funding
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Fulbright Foundation Scholar in Residence Program (Unknown)
Responsible Party: Principal Investigator, Michaela Kristina Farber, MD, Associate Professor, Harvard Medical School, Brigham and Women's Hospital
Other Study IDs: 2023P002364
Record Dates: First submitted 2023-10-11; First posted 2023-10-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Transthoracic Echocardiography; Antihypertensive Agents; Pregnancy
MeSH Terms: conditions — Pre-Eclampsia | interventions — Echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Preeclampsia: People with preeclampsia will be recruited at the time of diagnosis or suspected diagnosis of preeclampsia, according to accepted definitions of preeclampsia,2 nulliparous, singleton pregnancy, ≥ 20 weeks' gestation, without any preexisting cardiovascular, hepatic, or respiratory problems, no preexisting uterine abnormality including benign tumors, or placental adhesive disorder, not in labor, prior to treatment for preeclampsia, body mass index ≤ 40 kg/m2, age 18 to 50 years. Preeclampsia with severe features will be defined using the American College of Obstetrics and Gynecology definition
  Interventions: Diagnostic Test: Transthoracic Echocardiography
- Healthy Normotensive: Healthy pregnant people will be defined as American Society of Anesthesiologists (ASA) Classification II with no significant medical or surgical illness, nulliparous (first pregnancy beyond 20 weeks' gestation), non-smokers, singleton pregnancy with no uterine abnormalities and normally defined placentation. They will not be receiving any vasoactive medication including salbutamol or thyroid replacement hormones or have ruptured membranes.
  Interventions: Diagnostic Test: Transthoracic Echocardiography

INTERVENTIONS:
Diagnostic Test: Transthoracic Echocardiography — Cardiac output measured by transthoracic echocardiography (TTE)

SUMMARY:
The goal of this observational trial is to determine the resting cardiac output (CO) using transthoracic echocardiography (TTE) in a cohort of people with untreated preeclampsia, and a cohort of healthy normotensive pregnant people.

DETAILED DESCRIPTION:
This study seeks to evaluate cardiac output in people with untreated preeclampsia in a tertiary referral centre in the US. In doing so the investigators hope to better understand the underpinning of the pathophysiology of this condition and provide evidence for (or against) the new theory of the development of preeclampsia. The investigators also seek to examine CO changes at birth during cesarean delivery (CD) comparing healthy pregnant people with people with preeclampsia and further understand the changes in cardiac output (CO) after treatment with antihypertensive agents for preeclamptic patients so that the investigators may better rationale treatment with these agents and evaluate the changes that may occur at the time of CD and after cesarean birth in people with preeclampsia using TTE so that fluid therapy and blood pressure treatment can be prescribed based on hemodynamic findings. Further the investigators aim to imbed echocardiography into the management of people with preeclampsia and to determine the feasibility and long-term sustainability of conducting echocardiography studies in pregnant people with a multidisciplinary group at the Brigham and Women's Hospital Boston.

ELIGIBILITY:
Inclusion Criteria:

Preeclampsia Participant.

1. Preclampsia definition: People with preeclampsia will be recruited at the time of diagnosis or suspected diagnosis of preeclampsia, according to accepted definitions of preeclampsia. Preeclampsia with severe features will be defined using the American College of Obstetrics and Gynecology definition.
2. Nulliparous, singleton pregnancy,
3. ≥20 weeks gestation
4. without any preexisting cardiovascular, hepatic, or respiratory problems,
5. No preexisting uterine abnormality including benign tumors, or placental adhesive disorder,
6. Not in labor,
7. Not with prior to treatment for preeclampsia,
8. Body mass index ≤ 40 kg/m2, age 18 to 50 years.

Healthy Participant:

Healthy pregnant people will be defined as

1. American Society of Anesthesiologists (ASA) Classification II with no significant medical or surgical illness,
2. Nulliparous (first pregnancy beyond 20 week's gestation)
3. Non-smokers, singleton pregnancy
4. Not having ruptured membranes
5. No uterine abnormalities
6. No placentation abnormalities.
7. Not receiving any vasoactive medication including salbutamol
8. Not on thyroid replacement hormones

Exclusion Criteria:

Preeclampsia Participant:

1. Multiparous, multiple pregnancy,
2. Previous cardiovascular, hepatic or respiratory problems
3. Gestational diabetes,
4. Hemodynamic or neurologically unstable patient
5. Unable to tolerate a 30-minute ultrasound examination (TTE)
6. Age less than 18 or greater than 50 years
7. BMI > 40 kg/m2,
8. Gestation < 20 weeks.

Healthy Participant:

1. Current administration of vasoactive drugs including salbutamol
2. Current administration of thyroxine
3. Pre-existing or gestational diabetes
4. Tobacco use
5. Pre-existing or gestational hypertension or preeclampsia
6. Known uterine abnormality, in labor or ruptured membranes
7. Unable to tolerate a 30-minute ultrasound examination (TTE)
8. Age less than 18 or greater than 50 years
9. BMI > 40 kg/m2,
10. Gestation < 20 weeks.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant People
Study Population: 80 pregnant people will be recruited; 40 with preeclampsia, and 40 healthy normotensive pregnant people.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-10-25 (Estimated); Primary Completion 2027-10-11 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Cardiac output measured by transthoracic echocardiography (TTE) at rest: CO mL/min. | During gestation (8 wks to 42 wks, during clinic or hospital visits) with diagnosis of Preeclampsia
  Cardiac output measured by transthoracic echocardiography (TTE)

SECONDARY OUTCOMES:
cardiac output measured by transthoracic echocardiography (TTE) after treatment with antihypertensive agents, and during CD and postpartum | Post-treatment with antihypertensive (<60 min; during clinic or hospital ), Postpartum (cesarean or vaginal delivery; <60 min; immediately after to up to 6 hrs after delivery)
  Cardiac output measured by transthoracic echocardiography (TTE)

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Farber, MD, Principal Investigator — BWH; Alicia T Dennis, MBBS PhD MPH, Study Director — University of Melbourne, Australia
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Results may be the genesis of an international collaborative effort

REFERENCES:
- [Background] Dennis AT, Castro JM. Echocardiographic differences between preeclampsia and peripartum cardiomyopathy. Int J Obstet Anesth. 2014 Aug;23(3):260-6. doi: 10.1016/j.ijoa.2014.05.002. Epub 2014 May 29. PMID 24986564
- [Result] Dennis AT. Transthoracic echocardiography in women with preeclampsia. Curr Opin Anaesthesiol. 2015 Jun;28(3):254-60. doi: 10.1097/ACO.0000000000000182. PMID 25812006
- [Result] Dennis AT, Castro JM. Transthoracic echocardiography in women with treated severe pre-eclampsia. Anaesthesia. 2014 May;69(5):436-44. doi: 10.1111/anae.12623. Epub 2014 Mar 27. PMID 24673113